CLINICAL TRIAL: NCT05126030
Title: TRiCares Topaz Transfemoral Tricuspid Heart Valve Replacement System First in Human Trial
Brief Title: The TRICURE First in Human Trial
Acronym: TRICURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRiCares (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2101
Record Dates: First submitted 2021-10-28; First posted 2021-11-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Topaz TTVR System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Cohort (Experimental): Device: Topaz TTVR system
  Interventions: Device: Topaz TTVR System

INTERVENTIONS:
Device: Topaz TTVR System — Transcatheter tricuspid heart valve replacement

SUMMARY:
The objective of this first in human study is to gain early clinical insight into the safety profile and performance of the Topaz transcatheter tricuspid valve replacement (TTVR) system intended for transfemoral access to deliver a self-expanding bioprosthetic valve within the tricuspid valve.

DETAILED DESCRIPTION:
The TRiCares Topaz Prosthesis is intended to replace a diseased tricuspid heart valve via a transcatheter approach without removing the native valve.

ELIGIBILITY:
Inclusion Criteria:

* Subject of age >18 years.
* Subject with severe symptomatic tricuspid regurgitation presenting following conditions:

  1. TR severity of at least 3 (severe) on a scale of 0 (none) to 5 (torrential), assessed by independent core lab and/or
  2. symptoms requiring use of diuretics.
* Subject presenting with New York Heart Association Class NYHA ≥II.
* Subject is not eligible for open tricuspid valve surgery due to high operative risk, as determined by a Heart Team decision.

Exclusion Criteria:

* Subject in need of emergent or urgent intervention or any planned cardiac intervention within the next 12 months.
* Subject undergoing cardiac interventions within 30 days prior to index procedure.
* Subject with concomitant clinically relevant mitral, aortic, pulmonary regurgitation/stenosis.
* Subject who had previous tricuspid valve replacement or repair and a device is still in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite endpoint | 30 days
  including all-cause mortality, re-hospitalization for heart failure, re-intervention for failed tricuspid intervention, and KCCQ worsening at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Vanoverschelde, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Emmanuel Teiger, MD, Principal Investigator — CHU Henri Mondor
Locations (11):
- Belgium (4):
  - Algemeen Stedelijk Ziekenhuis,, Aalst
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc UCL, Brussels
  - Centre hospitalier universitaire CHU de Liège, Liège
- France (7):
  - CHU Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Hôpital Cardiothoracique Louis Pradel, Bron
  - CHU Henri Mondor, Créteil
  - University Hospital Lille, Institut Cœur Poumon, Lille
  - Hôpital Saint Joseph, Marseille
  - CHU Pontchaillou, Rennes
  - Centre Cardiologique du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teiger E, Nejjari M, Rosseel L, Kefer J, Verheye S, Lancellotti P, Oliver L, Obadia JF, Asch FM, Blanke P, Dreyfus J. TRICURE: first-in-human study of the Topaz transcatheter tricuspid heart valve system. EuroIntervention. 2025 Nov 14;21(22):1377-1385. doi: 10.4244/EIJ-D-25-00423. PMID 41243777